CLINICAL TRIAL: NCT02217540
Title: Mulligan Concept Mobilisation With Movement for Shoulder Dysfunction in Older Adults- A Pilot Randomised Clinical Trial
Brief Title: Mulligan Concept Mobilisation With Movement for Shoulder Dysfunction in Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alcala (Other)
Responsible Party: Principal Investigator, Cristina Lirio Romero, MSc. PhD student, University of Alcala
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Lirio-001-UAH
Record Dates: First submitted 2014-08-13; First posted 2014-08-15 (Estimated); Last update posted 2023-12-04 (Actual); Status verified 2014-08

CONDITIONS: Disorder of Shoulder
Keywords: Shoulder, disability evaluation, physiotherapy modalities
MeSH Terms: interventions — AIEOP acute lymphoblastic leukemia protocol; Movement

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Experimental Group (Experimental): Experimental Group consist of the physiotherapy standard protocol and active movement plus accessory mobilizations of the humeral head using Mulligan Concept Mobilisation with Movement.
  Interventions: Other: Standard protocol; Other: Mulligan Concept Mobilisation with Movement
- Control Group (Active Comparator): Standard protocol proposed by the Spanish Rheumatology Society for shoulder dysfunction
  Interventions: Other: Standard protocol

INTERVENTIONS:
Other: Standard protocol — Control group intervention is the physiotherapy treatment standard protocol proposed by the Spanish Rheumatology Society for shoulder dysfunction
  Other Names: Standard protocol for shoulder pain of Spanish Rheumatology Society
Other: Mulligan Concept Mobilisation with Movement — The internal hand of the physiotherapist stabilises participants´ shoulder girdle and with the thenar eminence of the other hand, performs a posterior-lateral glide of the humeral head. Participants are asked to raise the affected arm in the point of pain onset while the physiotherapist sustains the gliding force to humeral head. The physiotherapist tries to maintain the glide at right angles to the plane of movement throughout the entire range while participants are requested to perform an active elevation. Participants are instructed that the mobilisation procedure, including shoulder movement, had to be pain free
  Arms: Experimental Group

SUMMARY:
Objective: To pilot the methods proposed for conducting a full randomised clinical trial to evaluate the effect of Mulligan concept mobilization with movement on shoulder functionality in older adults with shoulder dysfunction.

Design: Pilot randomised, single-blinded clinical trial. Setting: Three nursing homes, Toledo, Spain. Participants: 44 older adults with shoulder dysfunction. Interventions: Participants will be randomly allocated into control group (n=22) treated with a physiotherapy standard protocol proposed by the Spanish Rheumatology Society; and experimental group (n=22) treated with the same physical therapy standard protocol and Mulligan concept mobilisation with movement. Both interventions will take place three times a week for 2 consecutive weeks.

Main outcomes: Primary outcome is shoulder functionality measured with Shoulder Disability Questionnaire (S-SDQ) Spanish version, and secondary outcomes are active glenohumeral range of motion and pain intensity. Data will be collected at baseline, after each group intervention, and 1 and 3 months after finishing interventions.

DETAILED DESCRIPTION:
Shoulder dysfunction is a common problem in older adults reaching up to 21% of prevalence. Shoulder symptoms, such as pain and reduced shoulder active range of motion (AROM) and function, might be associated to chronic pain, disability and decline in physical performance over time. Upper limbs and shoulder joint proper functionality leads to an adequate independence in activities of daily living (ADL) and functional performance. Therefore, maintaining independence in ADL and functional well-being in older adults should be a priority target for health care. A successful therapeutic approach depends on the understanding that the aging process is the responsible of major changes involving muscle disorders and joint stiffness.

Among the most common approaches to treating in¬dividuals with shoulder dysfunction, physiotherapy interven¬tion is often recommended as the first choice for a conservative treatment. Physiotherapy treatment usually includes therapeutic exercises, manual therapy, and various modalities and there are controversies about the most effective approach for pain reduc¬tion, increase in AROM and function, and decrease in disability in people with shoulder dysfunction. There is evidence about the effectiveness of thera¬peutic exercise, and the benefit of manual therapy for improvements in mobility and a trend in improving pain measures, while increases in function and quality of life are still questionable.

Some evidence was found about the effects of therapeutic exercise programs for overall performance improvement in older adults, but not specifically shoulder dysfunction. Regarding manual therapy in elderly, Knebl et al. developed a study about the effectiveness of Spencer manipulative technique in shoulder pain and found an improvement in functionality, shoulder AROM and pain intensity. Van den Dolder et al. investigated the effect of soft tissue massage on shoulder ROM, pain and dysfunction in patients with a mean age of 64 years old and found statistically significant results. Therefore, manual therapy techniques may be an option for correcting joint mechanics, promoting adhesion removal and restoring passive shoulder mobility in older adults.

Mobilisation with movement (MWM) is a manual therapy technique based on the analysis and correction of any minor positional fault in a joint. According to Mulligan, positional faults are due to various soft tissue and/or bone lesions in/around the joint and were explained in patients with shoulder pain by a kinematic study. This technique aims to realign joints positional faults by applying a manually specific oriented glide to a painful joint, assessing and adjusting force intensity, while the patient actively performs joint movement, so that patient's symptoms are immediately relieved and the maneuvers improve pain and movement. Therefore, when a correction mobilization is sustained, pain-free movement is restored and several repetitions are performed in order to get an improvement that lasts over time. The initial effects of MWM were assessed by Teys et al. in adults; who proved its effectiveness in increasing shoulder AROM and decreasing positional faults. Therefore, MWM may be an effective technique in physiotherapy treatment for shoulder dysfunction, as this it addresses passive and active shoulder structures. However, no studies about MWM effectiveness for shoulder dysfunction in older adults have been found.

The purpose of this pilot clinical trial is to pilot the methods proposed to conduct a full randomised controlled clinical trial to determine the effect of Mulligan concept MWM for shoulder dysfunction in older adults. The primary objectives are to evaluate the feasibility of recruitment, randomisation, retention, assessment procedures, and implementation of Mulligan concept MWM intervention. A secondary aim is to undertake a preliminary comparison of patient reported-outcomes and to estimate the variability of these outcomes in older adults with shoulder dysfunction.

ELIGIBILITY:
Inclusion Criteria:

* to be over 65 years old
* diagnosed with shoulder dysfunction (shoulder pain and/or limited AROM in the last 4 weeks) by their physician
* dependent on at least 1 ADL
* with a limited glenohumeral AROM of 25% - 75%
* resident in the nursing homes where the study took place.

Exclusion Criteria:

* subjects with moderate or severe cognitive impairment
* specific rheumatic diseases, osteoarthritis, neoplasms
* shoulder joint instability
* circulatory disorders (hemophilia, clotting problems)
* skin problems aggravated by contact with the skin
* traumas in the past month
* bilateral shoulder disorders

Ages: 65 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 44 (Actual)
Dates: Start 2012-01; Primary Completion 2013-01 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Spanish-Shoulder Disability Questionnaire | baseline and 3 times after interventions
  SDQ is mostly used in research and clinical practice in several countries and its score can range from minimum [0=no functional limitation] to maximum [100= affirmative to all items], so higher scores mean higher disability

SECONDARY OUTCOMES:
Range of motion and pain | baseline and 3 times after intervention
  glenohumeral range of motion (flexion, abduction, and external and internal rotations) measured with a universal goniometer (E Nonius-F®) and pain intensity measured with 11-point Verbal Numeric Rating Scale (VNS) for its good reliability and validity and usefulness in older adults

CONTACTS AND LOCATIONS:
Overall Officials: Cristina Lirio Romero, MsC, Principal Investigator — University of Alcala
Locations (1):
- Mensajeros de la Paz, Villarrubia de Santiago, Toledo, Spain

REFERENCES:
- [Background] Knebl JA, Shores JH, Gamber RG, Gray WT, Herron KM. Improving functional ability in the elderly via the Spencer technique, an osteopathic manipulative treatment: a randomized, controlled trial. J Am Osteopath Assoc. 2002 Jul;102(7):387-96. PMID 12138953
- [Background] van den Dolder PA, Roberts DL. A trial into the effectiveness of soft tissue massage in the treatment of shoulder pain. Aust J Physiother. 2003;49(3):183-8. doi: 10.1016/s0004-9514(14)60238-5. PMID 12952518
- [Background] Mulligan BR. Manual Therapy 'NAGS', 'SNAGS', 'MWMS' etc. 6 ed. Wellington: Orthopedic Physical Therapy Products; 2010
- [Background] Teys P, Bisset L, Vicenzino B. The initial effects of a Mulligan's mobilization with movement technique on range of movement and pressure pain threshold in pain-limited shoulders. Man Ther. 2008 Feb;13(1):37-42. doi: 10.1016/j.math.2006.07.011. Epub 2006 Oct 27. PMID 17070090
- [Result] Eggermont LH, Leveille SG, Shi L, Kiely DK, Shmerling RH, Jones RN, Guralnik JM, Bean JF. Pain characteristics associated with the onset of disability in older adults: the maintenance of balance, independent living, intellect, and zest in the Elderly Boston Study. J Am Geriatr Soc. 2014 Jun;62(6):1007-16. doi: 10.1111/jgs.12848. Epub 2014 May 13. PMID 24823985
- [Result] Chard MD, Hazleman R, Hazleman BL, King RH, Reiss BB. Shoulder disorders in the elderly: a community survey. Arthritis Rheum. 1991 Jun;34(6):766-9. doi: 10.1002/art.1780340619. PMID 2053923
- [Result] Vermeulen J, Neyens JC, van Rossum E, Spreeuwenberg MD, de Witte LP. Predicting ADL disability in community-dwelling elderly people using physical frailty indicators: a systematic review. BMC Geriatr. 2011 Jul 1;11:33. doi: 10.1186/1471-2318-11-33. PMID 21722355
- [Result] Koh ES, Jae-Young L. The management of shoulder pain in the elderly: focusing on clinical characteristics and conservative treatment. J Korean Geriatr Soc 2013;17(1):1-6
- [Result] Chester R, Shepstone L, Lewis JS, Jerosch-Herold C. Predicting response to physiotherapy treatment for musculoskeletal shoulder pain: protocol for a longitudinal cohort study. BMC Musculoskelet Disord. 2013 Jun 21;14:192. doi: 10.1186/1471-2474-14-192. PMID 23800352
- [Result] Brudvig TJ, Kulkarni H, Shah S. The effect of therapeutic exercise and mobilization on patients with shoulder dysfunction : a systematic review with meta-analysis. J Orthop Sports Phys Ther. 2011 Oct;41(10):734-48. doi: 10.2519/jospt.2011.3440. Epub 2011 Sep 4. PMID 21891875
- [Result] Camarinos J, Marinko L. Effectiveness of manual physical therapy for painful shoulder conditions: a systematic review. J Man Manip Ther. 2009;17(4):206-15. doi: 10.1179/106698109791352076. PMID 20140151
- [Result] de Vries NM, van Ravensberg CD, Hobbelen JS, Olde Rikkert MG, Staal JB, Nijhuis-van der Sanden MW. Effects of physical exercise therapy on mobility, physical functioning, physical activity and quality of life in community-dwelling older adults with impaired mobility, physical disability and/or multi-morbidity: a meta-analysis. Ageing Res Rev. 2012 Jan;11(1):136-49. doi: 10.1016/j.arr.2011.11.002. Epub 2011 Nov 11. PMID 22101330
- [Result] Chou CH, Hwang CL, Wu YT. Effect of exercise on physical function, daily living activities, and quality of life in the frail older adults: a meta-analysis. Arch Phys Med Rehabil. 2012 Feb;93(2):237-44. doi: 10.1016/j.apmr.2011.08.042. PMID 22289232
- [Result] Hurschler C, Wulker N, Mendila M. The effect of negative intraarticular pressure and rotator cuff force on glenohumeral translation during simulated active elevation. Clin Biomech (Bristol). 2000 Jun;15(5):306-14. doi: 10.1016/s0268-0033(99)00088-1. PMID 10758290
- [Result] Vicenzino B, Paungmali A, Teys P. Mulligan's mobilization-with-movement, positional faults and pain relief: current concepts from a critical review of literature. Man Ther. 2007 May;12(2):98-108. doi: 10.1016/j.math.2006.07.012. Epub 2006 Sep 7. PMID 16959529
- [Result] Ho CY, Sole G, Munn J. The effectiveness of manual therapy in the management of musculoskeletal disorders of the shoulder: a systematic review. Man Ther. 2009 Oct;14(5):463-74. doi: 10.1016/j.math.2009.03.008. Epub 2009 May 21. PMID 19467911
- [Result] Alvarez-Nemegyei J, Puerto-Ceballos I, Guzman-Hau W, Bassol-Perea A, Nuno-Gutierrez BL. Development of a Spanish-language version of the Shoulder Disability Questionnaire. J Clin Rheumatol. 2005 Aug;11(4):185-7. doi: 10.1097/01.rhu.0000173229.50674.31. PMID 16357754
- [Result] Jones KR, Fink R, Hutt E, Vojir C, Pepper GA, Scott-Cawiezell J, Mellis BK. Measuring pain intensity in nursing home residents. J Pain Symptom Manage. 2005 Dec;30(6):519-27. doi: 10.1016/j.jpainsymman.2005.05.020. PMID 16376738